CLINICAL TRIAL: NCT01574274
Title: Randomized Study of Intravenous Calaspargase Pegol (SC-PEG Asparaginase) and Intravenous Oncaspar in Children and Adolescents With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Brief Title: SC-PEG Asparaginase vs. Oncaspar in Pediatric Acute Lymphoblastic Leukemia (ALL) and Lymphoblastic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Shire (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew E. Place, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-001
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Results first posted 2022-09-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — calaspargase pegol; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SC-PEG (Arm A) (Active Comparator): Patients in this arm were randomized to receive IV Calaspargase Pegol (SC-PEG) 2500 IU/m2, administered as a single dose during induction and for 30 weeks post-induction. In the post-induction phases, IV SC-PEG was administered every 3 weeks (for a total of 10 post-induction doses). Protocol therapy was comprised of 5 phases: Induction, Consolidation I, CNS, Consolidation II, and Continuation, and varied based off risk classification.
  Interventions: Drug: SC-PEG
- Oncaspar (Arm B) (Active Comparator): Patients in this arm were randomized to receive IV Oncaspar 2500 IU/m2, administered as a single dose during induction and for 30 weeks post-induction. In the post-induction phases, IV Oncaspar was administered every 2 weeks (for a total of 15 post-induction doses). Protocol therapy was comprised of 5 phases: Induction, Consolidation I, CNS, Consolidation II, and Continuation, and varied based off risk classification.
  Interventions: Drug: Oncaspar

INTERVENTIONS:
Drug: SC-PEG — 11 doses Intravenously over one hour
  Arms: SC-PEG (Arm A)
Drug: Oncaspar — 16 doses Intravenously over one hour
  Arms: Oncaspar (Arm B)

SUMMARY:
This study is being conducted to learn about the effects of SC-PEG, which is a new form of a chemotherapy drug called asparaginase. Asparaginase is used to treat ALL and lymphoblastic lymphoma. The standard form of asparaginase, called Elspar, is given in the muscle once a week for 30 weeks. There are other forms of asparaginase. The investigators will be studying two of these: Oncaspar and Calaspargase Pegol (SC-PEG). The investigators have previously studied giving Oncaspar in the vein (instead of the muscle) every 2 weeks in patients with ALL, and have shown that this dosing did not lead to any more side effects than Elspar given weekly in the muscle. The study drug, SC-PEG, is very similar but not identical to Oncaspar. SC-PEG has been given in the vein to children and adolescents with ALL as part of other research studies, and it appears to last longer in the blood after a dose than Oncaspar. It has not yet been approved by the FDA. The goal of this research study is to learn whether the side effects and drug levels of SC-PEG given in the vein every 3 weeks are similar to Oncaspar given into the vein about every 2 weeks.

The study will also help to determine whether changing treatment for children and adolescents with ALL with high levels of minimal residual disease may improve cure rates. Measuring minimal disease (MRD) is a laboratory test that finds low levels of leukemia cells that the investigators cannot see under the microscope. In the past, it has been shown that children and adolescents with ALL with high levels of MRD after one month of treatment are less likely to be cured than those with low levels of MRD. Therefore, on the study, the bone marrow and blood at the end of the first month of treatment will be measured in participants with leukemia, and changes in therapy will be implemented based on this measurement. It is not known for sure that changing treatment will improve cure rates. MRD levels can only be measured if the marrow is filled with cancer cells at the time of diagnosis. Therefore, MRD studies will only be done in children and adolescents with ALL and not in those with lymphoblastic lymphoma.

Another part of the study is to determine whether giving antibiotics during the first month of treatment even to participants without fever will prevent serious infections in the blood and other parts of the body. About 25% of children and adolescents with ALL and lymphoblastic lymphoma who receive standard treatment develop a serious blood infection from a bacteria during the first month of treatment. Typically, antibiotics (medicines that fight bacteria) are given by vein only after a child with leukemia or lymphoma develops a fever or have other signs of infection. In this study, antibiotics will be given by mouth or in the vein to all participants during the first month of treatment, whether or not they develop fever.

Another goal of the study to learn how vitamin D levels relate to bone problems (such as broken bones or fractures) that children and adolescents with ALL and lymphoblastic lymphoma experience while on treatment. Some of the chemotherapy drugs used to treat ALL and lymphoblastic lymphoma can make bones weaker, which make fractures more likely. Vitamin D is a natural substance from food and sunlight that can help keep bones strong. The investigators will study how often participants have low levels of vitamin D while receiving chemotherapy, and, for those with low levels, whether giving vitamin D supplements will increase those levels.

Another focus of the study is to learn more about the biology of ALL and lymphoblastic lymphoma by doing research on blood, bone and spinal fluid bone marrow samples. The goal of this research is to improve treatment for children with leukemia in the future.

DETAILED DESCRIPTION:
To determine whether or not children and adolescents with ALL or lymphoblastic lymphoma are eligible to participate in this study, screening tests will be performed, which may include the following: medical history, bone marrow tests, assessment of your tumor, blood tests and/or an EKG.

Participants who enroll in this study will receive with anti-leukemia drugs called chemotherapy. During study treatment, the study doctors will continue to perform tests on blood, bone marrow and spinal fluid to assess how the disease is responding to the study treatment and to look for possible side effects. Scans (for example, x-ray, CT scan or MRI scan) may also be done after beginning study treatment to look for possible side effects. If the disease was initially diagnosed by a scan, it will also be repeated during the study treatment to assess how it is responding.

There are three different treatment groups in which leukemia and lymphoblastic lymphoma can be divided and they differ slightly in the types and amounts of chemotherapy drugs used during the 2-years of therapy. Participants are assigned to the different categories based on the features of their leukemia or lymphoma, such as their age, white blood cell count, and results of other tests. The three different treatment groups are called "Standard Risk", "High Risk" and "Very High Risk".

Participants will be given several different chemotherapy drugs during many periods of treatment (called "phases"). These drugs are known to kill lymphoblastic cancer cells. Some of the drugs are given by mouth, some into the veins (intravenously), and others as an injection (a shot) into the muscle. Some chemotherapy drugs will be given directly into your spinal fluid (called intrathecal chemotherapy) during a lumbar puncture (spinal tap). This treatment helps prevent the cancer cells from coming back in the spinal fluid and brain.

The first phase of treatment is steroid prophase. This phase of treatment is typically given in the hospital. This phase of treatment will begin immediately.

after enrolling on the study.

The second phase of treatment is remission induction. This phase will begin immediately after the steroid prophase and will last four weeks. Participants typically remain in the hospital for most (sometimes all) of this phase.

At the end of the remission induction phase, participants will undergo tests to determine if they are in remission. This testing will involve getting samples of blood, bone marrow and spinal fluid to look for cancer cells under the microscope. This testing will also involve getting repeat scans if these were not normal at the time of diagnosis. Remission means that cancer cells cannot be detected under the microscope in the blood, marrow and spinal fluid, and that any cancer previously seen on a scan has significantly improved or is no longer seen. Participants must be in remission to go onto the next phases of treatment; alternative treatments will be discussed with participants who are not in remission at the end of the induction phase.

The Consolidation I phase begins once it is determined that a participant is in remission. This phase lasts about three weeks. This phase of treatment is given in the hospital, but participants may be able to leave the hospital after the first week of the phase. The purpose of this phase is to further reduce the number of cancer cells in the body.

The next phase is the Central Nervous System (CNS) phase, and is usually given in the outpatient setting. Participants may need to be admitted to the hospital during this phase of treatment if a complication develops, such as infection. This phase of therapy begins immediately after the Consolidation I phase and lasts about 3 weeks. Treatment involves a series of lumbar punctures with anti-leukemia drugs given intrathecally over a two week period. Anti-leukemia drugs will also be given by mouth and by vein during this phase as well. Some participants may receive radiation therapy during this phase, although most do not. The decision to treat with radiation or not is based on characteristics of the cancer at diagnosis and whether or not cancer cells were seen in spinal fluid at that time. Radiation therapy is a painless procedure, the purpose of which is to prevent leukemia from coming back in the brain. For participants who receive radiation therapy, it will be given in either 8 or 10 daily treatments, depending on how many leukemia cells were seen in the spinal fluid under the microscope at diagnosis.

The next phase of the study is Consolidation II. This phase begins about 3 weeks after starting the CNS phase and lasts for about 27 weeks. During this phase, chemotherapy is given in three-week cycles, with some drugs given in clinic and some drugs given by mouth at home. Participants are typically treated as outpatients during this phase.

The last phase is called Continuation. This is also usually given as an outpatient. The goal of this phase is to rid the body of all remaining cancer cells. The cycles of chemotherapy during this phase are repeated every 3 weeks, with some drugs given in clinic and some drugs given by mouth at home. This phase will ends two years after remission was documented.

The randomization in this study involves the two forms of asparaginase, Oncaspar and SC-PEG asparaginase. Because no one knows which of the study options is best, participants will be "randomized" into one of the study groups: to receive Oncaspar or to receive SC-PEG. Randomization means that participants are put into a group by chance. Participants who are placed in the Oncaspar group will receive a single dose of Oncaspar on Day 7 of the Remission Induction phase, and then every 2 weeks for 30 weeks starting in the CNS phase (16 total doses of Oncaspar). Participants placed in the SC-PEG group will receive SC-PEG asparaginase on Day 7 of the remission induction phase and then every 3 weeks beginning in the CNS phase (11 total doses of SC-PEG).

Minimal Residual Disease (MRD) testing is a way to look for very low levels of leukemia in the body that cannot be seen under the microscope. These test will be done in a laboratory at Dana-Farber Cancer Institute. If the MRD results are in the low range on Day 32, thre will be no change to the treatment program described above. If the MRD results are in the high range, then it will be recommended that treatment be changed.

Participants will receive a fluoroquinolone antibiotic beginning during the first phase of treatment and continuing until the neutrophils and monocytes (two types of white blood cells in the blood that help fight infection) have increased. The goal of giving the antibiotics is to prevent infection during the first few weeks of treatment.

Participants who agree to have extra blood drawn to test for vitamin D levels in the blood will have 1 teaspoon of blood drawn at the following times: start of treatment, at the end of the first month of treatment, at the start of the continuation phase, and at the end of treatment. Participants will receive the results of these tests. If the vitamin D level is low, the study doctor will recommend that the participant take a vitamin D supplement. Participants may choose not to have blood drawn to check vitamin D levels, or may choose not to take the vitamin D supplement.

Participants will be asked at the time of study entry if they agree to provide additional blood and bone marrow samples for research. These additional samples will be used to learn more about the biology of ALL and lymphoblastic lymphoma. Stored specimens may also be used for future research regarding leukemia.

After completing all treatment, participants will be asked to come in for physical exams and blood work every month for the first six months after the final treatment, then every two months for the next 6 months, then every four months for the next year, and then every six months for the next year. After that we will ask you to come in once a year.

The investigators would like to keep track of the medical condition of all participants for the rest of their lives. This will be done by reviewing medical records of participants. The investigators may telephone participants who have finished treatment to see how they are doing if they have not been seen by their doctor for at least a year.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ALL or lymphoblastic leukemia
* No prior therapy except short courses of corticosteroids, a single dose of IT cytarabine or emergent radiation to the mediastinum or other life-threatening masses

Exclusion Criteria:

* Have received more than 7 days of corticosteroids in the preceding 4 weeks or more than 28 days of corticosteroids in the preceding 6 months
* Have received any chemotherapy or radiotherapy for previous malignancy
* Receiving any other investigational agent
* Known to be HIV positive
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding
* History of previous malignancy

Ages: 365 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2012-06; Primary Completion 2021-07 (Actual); Study Completion 2027-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Place, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (5):
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Montefiore Medical Center, New York, New York
  - Hasbro Children's Hospital, Providence, Rhode Island
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Hospital Sainte Justine, University of Montreal, Montreal, Quebec
  - Centre Hospitalier U. de Quebec, Québec, Quebec

REFERENCES:
- [Result] Vrooman LM, Blonquist TM, Stevenson KE, Supko JG, Hunt SK, Cronholm SM, Koch V, Kay-Green S, Athale UH, Clavell LA, Cole PD, Harris MH, Kelly KM, Laverdiere C, Leclerc JM, Michon B, Place AE, Schorin MA, Welch JJG, Neuberg DS, Sallan SE, Silverman LB. Efficacy and Toxicity of Pegaspargase and Calaspargase Pegol in Childhood Acute Lymphoblastic Leukemia: Results of DFCI 11-001. J Clin Oncol. 2021 Nov 1;39(31):3496-3505. doi: 10.1200/JCO.20.03692. Epub 2021 Jul 6. PMID 34228505
- [Derived] Cole PD, Kim SY, Li Y, Schembri A, Kelly KM, Sulis ML, Vrooman L, Welch JJG, Ramjan S, Silverman LB, Sands SA. Feasibility of serial neurocognitive assessment using Cogstate during and after therapy for childhood leukemia. Support Care Cancer. 2023 Jan 10;31(2):109. doi: 10.1007/s00520-022-07566-6. PMID 36625831
- [Derived] Burns MA, Place AE, Stevenson KE, Gutierrez A, Forrest S, Pikman Y, Vrooman LM, Harris MH, Hunt SK, O'Brien JE, Asselin BL, Athale UH, Clavell LA, Cole PD, Gennarini LM, Kahn JM, Kelly KM, Laverdiere C, Leclerc JM, Michon B, Schorin MA, Sulis ML, Welch JJG, Neuberg DS, Sallan SE, Silverman LB. Identification of prognostic factors in childhood T-cell acute lymphoblastic leukemia: Results from DFCI ALL Consortium Protocols 05-001 and 11-001. Pediatr Blood Cancer. 2021 Jan;68(1):e28719. doi: 10.1002/pbc.28719. Epub 2020 Oct 7. PMID 33026184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from June 3, 2012 to June 8, 2015.
Groups:
- SC-PEG (Arm A): Patients in this arm were randomized to receive IV Calaspargase Pegol (SC-PEG) 2500 IU/m2, administered as a single dose during induction and for 30 weeks post-induction. In the post-induction phases, IV SC-PEG was administered every 3 weeks (for a total of 10 post-induction doses). Protocol therapy was comprised of 5 phases: Induction, Consolidation I, Central Nervous System (CNS), Consolidation II, and Continuation, and varied based off risk classification.
Period: Overall Study
Arm/Group | SC-PEG (Arm A) | Oncaspar (Arm B)
Started (Randomized) | 119 | 121
Evaluable for Induction Events | 115 | 115
Achieved Complete Remission | 109 | 114
Received Post-induction Asparaginase | 109 | 114
Eligible | 119 | 120
Completed | 87 | 99
Not Completed | 32 | 22
Not completed — Ineligible | 0 | 1
Not completed — Withdrawal of Consent During Induction | 1 | 1
Not completed — Ph+ B-ALL | 3 | 4
Not completed — Induction Death | 2 | 0
Not completed — Induction Failure | 4 | 1
Not completed — Adverse Event | 16 | 13
Not completed — Remission Death | 1 | 0
Not completed — Withdrawal from Treatment but Agrees to be Followed | 2 | 0
Not completed — Other, unknown | 3 | 2

BASELINE CHARACTERISTICS:
Population: This analysis dataset is comprised of all eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | SC-PEG (Arm A) | Oncaspar (Arm B) | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Customized [Count of Participants; unit: Participants]
  < 10 years old | 89 | 90 | 179
  >/= 10 years old | 30 | 30 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 49 | 92
  Male | 76 | 71 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 74 | 77 | 151
  Unknown or Not Reported | 33 | 29 | 62
Immunophenotype [Count of Participants; unit: Participants]
  B-immunophenotype | 103 | 104 | 207
  T-immunophenotype | 16 | 16 | 32
Initial Dana-Farber Cancer Institute (DFCI) risk group [Count of Participants; unit: Participants] — Standard Risk (all of the following): Age 1-10 years, WBC < 50,000/microliter, B-ALL, CNS-1 or CNS-2.
  High Risk (any of the following): Age >=10 years, WBC >= 50,000/microliter, T-ALL, CNS-3.
  Participants
    Standard Risk | 70 | 71 | 141
    High Risk | 49 | 49 | 98
White Blood Cell (WBC) at diagnosis (cells/uL) [Count of Participants; unit: Participants]
  < 50,000 | 93 | 96 | 189
  >/= 50,000 | 21 | 20 | 41
  Missing | 5 | 4 | 9
CNS status at diagnosis [Count of Participants; unit: Participants] — CNS-1: no blast cells in cytospin, regardless of cerebrospinal fluid (CSF) cell count.
  CNS-2: Fewer than 5 white blood cell (WBC) on CSF cell count, with blasts on cytospin.
  CNS-3: 5 or more WBC on CSF cell count, with blasts on cytospin. Traumatic tap: > 10 red blood cell (RBC) on CSF cell count.
  Participants
    CNS 1 | 90 | 99 | 189
    CNS 2 | 19 | 15 | 34
    CNS 3 | 1 | 3 | 4
    Traumatic with Blasts | 3 | 2 | 5
    Traumatic without Blasts | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Asparaginase-Related Toxicity
Description: Asparaginase-related toxicity rate is defined as the percentage of patients who experience allergy (all grades), symptomatic pancreatitis (grade 2 or worse), thrombotic or bleeding complications requiring intervention (grade 2 or worse) with treatment attribution of possibly, probably or definite based on Common Terminology Criteria for Adverse Events (CTCAE) v4.
Time Frame: 30-week post-induction asparaginase treatment period. Toxicities assessed on an ongoing basis (at least 1 per month) while participant is on study, an average of 2 years.
Population: The analysis dataset is comprised of all patients who received post-induction asparaginase.
Measure: Count of Participants; unit: Participants
Arm/Group | SC-PEG (Arm A) | Oncaspar (Arm B)
Number analyzed (Participants) | 109 | 114
Participants | 41 | 43
Statistical Analysis 1: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Test type: Superiority; p = 1.00, Fisher Exact

2. Primary Outcome: Induction and Post-Induction Nadir Serum Asparaginase Activity Level
Description: Nadir serum asparaginase activity (NSAA) levels were estimated based on established methods.
Time Frame: Samples for nadir serum asparaginase activity levels were assayed at 4,11,18,and 25 days after 1st dose, and then prior to asparaginase dose given during post-induction, at Week 7, 13, 19, and 25.
Population: The analysis dataset is comprised of all randomized patients who consented to research studies with an evaluable sample for analysis of serum asparaginase activity at the respective induction and post-induction assessment timepoints.
Measure: Median (Full Range); unit: IU/mL
Arm/Group | SC-PEG (Arm A) | Oncaspar (Arm B)
Number analyzed (Participants) | 119 | 120
IU/mL
  Day 4 NSAA Level: number analyzed (Participants) | 77 | 79
  Day 4 NSAA Level | 0.975 [0.430 to 1.499] | 1.045 [0.069 to 1.731]
  Day 11 NSAA Level: number analyzed (Participants) | 60 | 60
  Day 11 NSAA Level | 0.571 [0.156 to 1.176] | 0.673 [0.025 to 1.224]
  Day 18 NSAA Level: number analyzed (Participants) | 62 | 60
  Day 18 NSAA Level | 0.394 [0.080 to 0.887] | 0.314 [0.025 to 0.536]
  Day 25 NSAA Level: number analyzed (Participants) | 42 | 47
  Day 25 NSAA Level | 0.319 [0.025 to 0.549] | 0.056 [0.025 to 0.079]
  Week 7 NSAA Level | 1.006 [0.025 to 1.948] | 1.097 [0.506 to 1.814]
  Week 13 NSAA Level | 1.147 [0.143 to 2.181] | 1.101 [0.512 to 1.866]
  Week 19 NSAA Level | 1.110 [0.318 to 2.709] | 1.134 [0.508 to 1.820]
  Week 25 NSAA Level | 1.117 [0.153 to 2.106] | 1.109 [0.483 to 1.814]
Statistical Analysis 1: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Day 4 NSAA Level; Test type: Superiority; p = 0.07, t-test, 2 sided
Statistical Analysis 2: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Day 11 NSAA Level; Test type: Superiority; p = 0.29, t-test, 2 sided
Statistical Analysis 3: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Day 18 NSAA Level; Test type: Superiority; p = 0.0002, t-test, 2 sided
Statistical Analysis 4: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Day 25 NSAA Level; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Week 7 NSAA Level; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Week 13 NSAA Level; Test type: Superiority; p = 0.87, t-test, 2 sided
Statistical Analysis 7: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Week 19 NSAA Level; Test type: Superiority; p = 0.83, t-test, 2 sided
Statistical Analysis 8: Comparison: SC-PEG (Arm A) vs Oncaspar (Arm B); Week 25 NSAA Level; Test type: Superiority; p = 0.94, t-test, 2 sided

3. Secondary Outcome: Frequency of Infections
Description: Number of episodes of bacteremia, fungemia and invasive fungal infections during the remission induction phase
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Outcome
Description: Rates of complete remission, relapse, induction death, remission death, and second malignant neoplasms in participants
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Outcome of Participants With Very-high Risk Disease
Description: Rates of relapse, remission death and second malignant neoplasm in participants with high minimal residual disease (MRD) and/or high risk cytogenetics who are treated with a more intensified regimen
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Feasibility of Vitamin D Screening/Supplementation
Description: Vitamin D-levels at various times during treatment, proportion of participants with low vitamin D levels, proportion of participants who agree to Vitamin D supplementation
Time Frame: 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Feasibility of Prospective Screening for ABGD
Description: Number of samples from participants with T-ALL in which a successful result was obtained by quantitative polymerase chain reaction (qPCR) to assess absence of biallelic TCRy deletions (ABGD); frequency of ABGD in T-ALL
Time Frame: 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Feasibility of Prospective Screening for Genetic Abnormalities
Description: Number of samples from participants with B-ALL in which a successful result was obtained in prospective screening for abnormalities (eg, mutations, deletions, rearrangements) of IKZF1, CRLF2 and JAK1/2 in patients with newly diagnosed B-ALL; proportion of participants with B-ALL found to have one of these abnormalities.
Time Frame: 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Relationship Between Apoptotic/Anti-apoptotic Proteins and Response to CT
Description: Levels of pro- and anti-apoptotic proteins in participant samples from diagnosis; correlation of these levels to clinical response (induction failure, high MRD, relapse).
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were continuously monitored and recorded prior to each course of therapy, for the duration of prophase, induction, and the total planned post-induction treatment of 24 months from complete remission (CR) date. Treatment duration for this study cohort was a median (range) of 769 days (3-797 days). AE assessment was performed at least 1x per month through the end of the Consolidation II phase, and at least 1x per 3 months during the Continuation phase, for a max of 797 days.
Description: AEs were collected by grade and treatment attribution, and max grade by toxicity type was calculated. Serious AEs were identified separately, and were defined as any adverse drug experience that resulted in any of the following: death, a life-threatening event, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. All remaining adverse events, regardless of attribution, were classified as Other AEs.
Arm/Group | SC-PEG (Arm A) | Oncaspar (Arm B)
All-Cause Mortality (participants affected / at risk) | 7/119 | 5/120
Serious Adverse Events (participants affected / at risk) | 35/119 | 27/120
Other Adverse Events (participants affected / at risk) | 118/119 | 120/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SC-PEG (Arm A) (N=119) | Oncaspar (Arm B) (N=120)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 10 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Edema trunk (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 4 | 1
Lung infection (Infections and infestations) | 3 | 1
Pleural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 9
Upper respiratory infection (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 5 | 2
Creatinine increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 6 | 12
Serum amylase increased (Investigations) | 3 | 5
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SC-PEG (Arm A) (N=119) | Oncaspar (Arm B) (N=120)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 55 | 57
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Anal mucositis (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 2
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 2
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 33 | 24
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 14 | 15
Rectal mucositis (Gastrointestinal disorders) | 0 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 1
Typhlitis (Gastrointestinal disorders) | 9 | 3
Edema limbs (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 2
Infusion site extravasation (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Irritability (General disorders) | 0 | 1
Localized edema (General disorders) | 2 | 0
Pain (General disorders) | 0 | 2
Fever (General disorders) | 0 | 1
Localized edema (General disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 17 | 15
Anaphylaxis (Immune system disorders) | 2 | 3
Abdominal infection (Infections and infestations) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0
Bone infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 3 | 7
Device related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 3
Hepatic infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 32 | 33
Lip infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 6 | 7
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 0 | 3
Skin infection (Infections and infestations) | 3 | 5
Soft tissue infection (Infections and infestations) | 3 | 1
Splenic infection (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Fracture (Injury, poisoning and procedural complications) | 19 | 20
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 4 | 7
Activated partial thromboplastin time prolonged (Investigations) | 15 | 18
Alanine aminotransferase increased (Investigations) | 100 | 98
Alkaline phosphatase increased (Investigations) | 12 | 8
Aspartate aminotransferase increased (Investigations) | 71 | 76
Blood bilirubin increased (Investigations) | 63 | 62
CPK increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 3 | 3
Ejection fraction decreased (Investigations) | 0 | 1
Fibrinogen decreased (Investigations) | 26 | 33
GGT increased (Investigations) | 3 | 0
INR increased (Investigations) | 14 | 8
Investigations - Other, specify (Investigations) | 2 | 1
Lipase increased (Investigations) | 23 | 23
Serum amylase increased (Investigations) | 27 | 22
Weight gain (Investigations) | 2 | 0
Weight loss (Investigations) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Glucose intolerance (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 53 | 47
Hyperkalemia (Metabolism and nutrition disorders) | 13 | 21
Hypernatremia (Metabolism and nutrition disorders) | 3 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 37 | 44
Hypoalbuminemia (Metabolism and nutrition disorders) | 98 | 102
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 41 | 46
Hypokalemia (Metabolism and nutrition disorders) | 63 | 54
Hyponatremia (Metabolism and nutrition disorders) | 29 | 28
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 9 | 12
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 7 | 1
Stroke (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 5
Vasovagal reaction (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal calculi (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 21 | 22
Hypotension (Vascular disorders) | 4 | 6
Thromboembolic event (Vascular disorders) | 20 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT01574274/Prot_SAP_000.pdf